CLINICAL TRIAL: NCT06312774
Title: Feasibility Study for Comparative Analysis of Proteome and Single-cell RNA Sequencing in Chronic Lung Disease Patients With and Without Sarcopenia
Brief Title: Feasibility of Proteomics in Chronic Lung Disease With Sarcopenia
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 333853
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Sarcopenia; Chronic Lung Disease
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Chronic Lung Disease
  Interventions: Other: This is observational study
- Healthy Controls
  Interventions: Other: This is observational study

INTERVENTIONS:
Other: This is observational study — This is observational study

SUMMARY:
Sarcopenia, the loss of muscle mass and strength with ageing, is a prevalent condition in older adults, particularly those with chronic lung diseases like COPD and interstitial lung disease. The condition exacerbates the decline in physical ability, leading to decreased mobility, impaired quality of life, and increased disability. Sarcopenia's prevalence varies across populations, estimated to affect up to 10% of adults over 60 worldwide, with higher rates reported in studies employing consensus definitions of sarcopenia. The prevalence is even higher in patients with chronic lung diseases, reaching up to 26.6%. Sarcopenia's impact on health-related quality of life has been widely investigated. The condition is associated with various comorbidities, including chronic heart failure, obesity, diabetes, and chronic kidney disease, all negatively impacting the quality of life.

The proposed study's primary aim is to assess the feasibility of the FACS (finding, assessing, confirming, severity) approach in determining sarcopenia's prevalence in the chronic lung disease population. FACS includes screening, strength measurements, and bioelectrical impedance analysis (BIA) to confirm sarcopenia.

The study will also explore potential mechanisms associated with sarcopenia in this population, using proteome and single-cell transcriptome profiles. These multi-omics approaches provide a comprehensive view of the cellular and molecular changes underlying sarcopenia.In particular, the study will evaluate patient acceptance, time efficiency of each test, and recruitment effectiveness. The outcomes will guide the design and execution of subsequent, larger studies and provide preliminary data for power calculation for the full-scale study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients diagnosed with chronic lung disease (≥ 18years).
2. Only patients who are willing and able to provide informed consent to participate in the study.

Exclusion Criteria:

1. Patients with other major comorbidities that could significantly impact muscle mass and function, such as severe heart failure, advanced liver or kidney disease, uncontrolled diabetes, or malignancies.
2. Patients with acute exacerbations of their chronic lung disease or any other acute illness at the time of the study. 3. Patients with a history of neuromuscular disorders or disability that could significantly affect muscle mass and function.

4. Patients who have undergone recent surgery in the past 6 months or have received specific treatments that could influence muscle mass and function, such as long-term corticosteroid use, chemotherapy, or radiation therapy.

5. Patients with life expectancy of less than 6 months 6. Patients who are unable or unwilling to comply with the study protocol or procedures.

7. Patients that are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sarcopenia, the condition of losing muscle mass and strength as we age, is especially common in older adults who also have chronic lung diseases such as COPD (a type of obstructive lung disease that makes it hard to breathe) and interstitial lung disease (a type of lung disease that affects the tissue and space around the air sacs of the lungs).
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2024-04-18 (Estimated); Primary Completion 2025-11-07 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia | 3 years
  feasibility of using the FACS approach and molecular analyses to investigate the association between sarcopenia and chronic lung disease